CLINICAL TRIAL: NCT06247293
Title: A Retrospective Study of Surgical Resection Combined With Intraperitoneal Hyperthermic Chemotherapy in the Treatment of Ruptured Hepatocellular Carcinoma
Brief Title: Surgical Resection Combined With Intraperitoneal Hyperthermic Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-KY-078-02
Record Dates: First submitted 2023-08-11; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-06

CONDITIONS: Hyperthermic Intraperitoneal Chemotherapy; Hepatocellular Carcinoma; Ruptured Liver
Keywords: ruptured and bleeding of Hepatocellular carcinoma; Hyperthermic intraperitoneal chemotherapy; recurrence-free survival
MeSH Terms: conditions — Carcinoma, Hepatocellular; Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Surgical resection combined with intraperitoneal hyperthermic perfusion chemotherapy: Surgical resection combined with intraperitoneal hyperthermic perfusion chemotherapy
  Interventions: Procedure: intraperitoneal hyperthermic perfusion chemotherapy
- simple surgical resection: Control group: simple surgical resection
  Interventions: Procedure: intraperitoneal hyperthermic perfusion chemotherapy
- other: imple interventional hemostasis group
  Interventions: Procedure: intraperitoneal hyperthermic perfusion chemotherapy

INTERVENTIONS:
Procedure: intraperitoneal hyperthermic perfusion chemotherapy — （1）Partial hepatectomy: The reasonable resection method was selected according to the tumor location, residual liver volume and the operation process. The tumor margin should be more than 1 cm, the abdominal cavity was flushed with sterile warm distilled water. In the control group,1-2 abdominal drainage tubes were placed on the hepatic cross-section, in the exposed group,4 abdominal perfusion tubes were placed in the right hepatic apex, splenic fossa, left and right pelvic cavity to perform HIPEC postoperatively.
  (2) HIPEC: Temperature setting:43 °C perfusion time:60 min, perfusion speed:400-600 mL/min ,perfusion volume:3000 mL.
  （3）Hepatic artery embolization：Through the common femoral artery, the catheter passed through the abdominal aorta, celiac trunk, the common hepatic artery and the inherent hepatic artery to the blood supply target artery of liver cancer. The embolic agent Lipiodol was mixed and injected to embolize the bleeding artery to stop bleeding.
  Other Names: simple surgical resection; Hepatic artery embolization

SUMMARY:
Patients with ruptured liver cancer and bleeding after surgical resection were included according to the criteria of admission, and the patients were divided into experimental and control groups. the primary efficacy end point was RFS, and the secondary end point was the rate of abdominal implant metastases and OS.To analyze the efficacy of HIPEC.

DETAILED DESCRIPTION:
Patients with ruptured liver cancer and bleeding after surgical resection were included according to the criteria of admission, and the patients were divided into groups: experimental group: surgical resection combined with intraperitoneal hyperthermic perfusion chemotherapy, and control group: simple surgical resection.

At further follow-up, the primary efficacy end point was time to Recurrence free survival (RFS) ,the time from the patient's treatment until the discovery of abdominal metastases or until the follow-up period, and the secondary end point was the rate of abdominal implant metastases, that is, according to the postoperative follow-up test and imaging findings, the incidence of abdominal implantation and metastasis, until the end of abdominal recurrence or metastasis or observation period. Overall Survival OS and survival rate: the time from the time the patient underwent partial hepatectomy until death from tumor causes or the end of the observation period. To analyze the efficacy of HIPEC.

ELIGIBILITY:
Inclusion Criteria:

1. according to the clinical diagnostic criteria of primary liver cancer (2022 edition) or confirmed by pathology/cytology;
2. preoperative diagnosis of rupture and hemorrhage of liver cancer by clinical manifestation, examination and imaging;
3. Age 18-80 years;
4. Child-pugh class A or class B after liver protection and albumin correction, without severe heart, lung or renal dysfunction, without absolute contraindication to surgery;
5. ECOG-PS score of 0-1;
6. without other neoplastic diseases;
7. Sign and perfect the informed consent form before operation;
8. without postoperative liver failure, without major complications such as massive hemorrhage, purulent infection and multiple organ failure, and without discharge from hospital.

Exclusion Criteria:

1. having other active malignant tumor;
2. the expected survival time is less than 3 months;
3. Child-pugh class C, complicated with severe organic disease of important organs, complicated with severe cirrhosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From February 2017 to February 2023, patients with ruptured Southern Medical University of hepatocellular carcinoma diagnosed in the Department of Hepatobiliary Surgery of Pearl River Hospital or other hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-02-25 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Intra-abdominal recurrence-free survival (RFS) | the time from surgical resection in patients with HCC until the detection of intra-abdominal recurrence or metastasis or the end of the observation period(2 years)
  Intra-abdominal recurrence-free survival (RFS):the time from surgical resection patients with HCC until the detection of intra-abdominal recurrence or metastasis or the end of the observation period, based on postoperative follow-up test criteria and imaging findings(2 years)

SECONDARY OUTCOMES:
Overall Survival (OS) | time from partial hepatectomy for HCC until death from any cause or end of observation period(2 years)
  Overall Survival (OS): time from partial hepatectomy for HCC until death from any cause or end of observation period(2 years)
survival rate | time from partial hepatectomy for HCC until death from any cause or end of observation period
  defined as 1-month,3-month,6-month, 1-year,2-year survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Mingxin Pan, Prof., Principal Investigator — Southern Medical University, China